CLINICAL TRIAL: NCT05870046
Title: Effectiveness of Power Training Compared With Non-specific Exercises on Functionality and Body Composition in Women Older Than 65 Years With Probable Sarcopenia.
Brief Title: Effectiveness of Power Training in Older Women With Pre-sarcopenia
Acronym: POSARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Luis Polo Ferrero, Associate Professor, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USalamancaPowerSarcopenia
Record Dates: First submitted 2023-05-08; First posted 2023-05-23 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Pre-sarcopenia; Old Age; Debility
Keywords: exercise; elderly; resistance training; sarcopenia
MeSH Terms: conditions — Frailty; Motor Activity; Sarcopenia

STUDY DESIGN:
Intervention Model Description: Longitudinal prospective, controlled, single-blind study
Who Masked: Participant, Outcomes Assessor
Masking Description: Single blind masking with blinded assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- power exercise group (Experimental): The main part of the muscle power exercise program will have the following exercises: wall push-ups, arm raises, elbow push-ups and extensions, weighted pronosupination, hand press, knee and hip hinge squat, dead weight, front and sagittal plan stride, and heel raises.
  It will have different phases:
  * 1st phase: exercise adaptation: the correct execution of upper and lower limb exercises will be taught for one month.
  * 2nd phase: Resistance training: During the following two months, strength exercises will be performed at slow and normal speed of the movement patterns learned in the training course.
  * 3rd phase: Muscle power training: During the last five months. A correct progression of the load and a progressive increase in the speed of execution of the different exercises will be carried out, gradually increasing the levels of difficulty and intensity.
  Interventions: Procedure: Power training in women older than 65 years with pre-sarcopenia
- multimodal exercise group (Active Comparator): The main part of the multicomponent exercise program integrates different exercise modalities: Aerobic, mobility, strength, balance and coordination exercises, playful activities or games are also included with some activities aimed at working on cognitive functions to reinforce the overall effects of the program, such as games with colors, numbers, letters, right-left laterality, memory, etc.
  The progression of the different models is as follows:
  * E. Aerobic: Start with continuous work, then intervallic, and decrease rest times in intervallic work.
  * E. Strength: Increase sets, repetitions and decrease rest time.
  * Balance: start with static and evolve with blindfolds, perturbations, dynamic balance, etc.
  * Coordination, and cognitive games will also become more complicated, with more complicated and faster decision making.
  Interventions: Procedure: Multimodal and nonspecific exercises in women older than 65 years with pre-sarcopenia
- Control group (No Intervention): Participants in this group should continue with their usual dietary pattern and level of physical activity, without changing their lifestyle habits during the study period. They will not participate in the strength exercise program based on muscle power, nor will they perform systematic, programmed and supervised physical exercise in any other program.

INTERVENTIONS:
Procedure: Power training in women older than 65 years with pre-sarcopenia — resistance training based on muscle power training, perform the exercises at high speed.
  Arms: power exercise group
Procedure: Multimodal and nonspecific exercises in women older than 65 years with pre-sarcopenia — different exercise modalities are integrated: Aerobic, mobility, strength, balance and coordination exercises.
  Arms: multimodal exercise group

SUMMARY:
This is a randomized, parallel, double-blind clinical trial. The main objective is to compare the efficacy of resistance training based on power training, multimodal exercise with non-specific exercises and a control group on functionality and body composition in women over 65 years of age with pre-sarcopenia.

The intervention in both groups will be carried out for 30 weeks, with three weekly sessions. Two evaluations will be performed, one pre-intervention and one post-intervention. Functionality (Timed Up & Go test (TUG), chair stand test and hand grip test and Short Physical Performance Battery (SPPB)), body composition (Body fat %, skeletal muscle index (SMI), appendicular skeletal muscle (ASM), waist circumference, waist hip ratio, body weight, body mass index (BMI)) will be evaluated.

DETAILED DESCRIPTION:
Design: Randomized, controlled clinical trial with three parallel groups, in which women over 65 years of age will be recruited. Study participants will be assigned to one of the three interventions. The study will have a duration of 8 months. There will be 2 evaluation visits, an initial one, a final one at 8 months. During 8 months there will be 3 weekly sessions lasting 50 minutes.

Scope: The study will be carried out in the Salamanca Health Area, in collaboration with the Research, Teaching and Assistance Unit of the Faculty of Nursing and Physiotherapy of the University of Salamanca and the Department of Elderly People of the Salamanca City Council.

Interventions: 1) Multimodal Exercise Group (GEM); 2) Muscle Power Exercise Group (GEP); 3) No Exercise Control Group (CG). The GEM and GEP sessions follow the same structural pattern. They will be structured according to the recommendations of the American College of Sports Medicine (ACSM). In the main part of the GEP, strength exercises will be performed and the speed will be progressively increased until the exercises are performed at the maximum speed that each participant can do.

Study population: 104 subjects over 65 years of age from the city of Salamanca will be included, distributed in 3 groups at a 1:1:1 ratio. Randomization will be performed using the Epidat 4.2 program. The sample size was calculated using GRANMO Version 7. 12 April 2012.

The main study variables are: Functionality (Timed Up & Go test (TUG), chair stand test and hand grip test and Short Physical Performance Battery (SPPB)), body composition (Body fat %, skeletal muscle index (SMI), appendicular skeletal muscle (ASM), waist circumference, waist hip ratio, body weight, body mass index (BMI)), SARC-F Questionnaire, % RM estimated by force-velocity profile and Gait speed.

Population characteristics will be presented as mean and standard deviation for continuous variables and as frequency distribution for qualitative variables. Statistical analysis The effect of the intervention on the study variables if the variables are parametric, Student's t-test will be used, and if they are non-parametric, the Wilcoxon test will be used. An alpha risk of 0.05 is set as the limit of statistical significance. The statistical program to be used will be SPSS, v.26.0.

The study will be carried out with the authorization of the Ethics Committee on Drug Research (CEIm) of the Salamanca Health Area, and with the prior informed consent of the study subjects. The participants will be informed of the objectives of the project and of the risks and benefits of the examinations and interventions to be performed. The study has been designed and subsequently assessed in accordance with Law 14/2007 on Biomedical Research, the ethical principles of the Declaration of Helsinki of the World Medical Association on ethical principles for medical research involving human subjects, as well as the other ethical principles and legal regulations applicable according to the characteristics of the study.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 65 years.
* pre-sarcopenia state (chair stand test > 15s or Hand Grip Strength < 16Kg).

Exclusion Criteria:

* Tumors
* Pacemakers
* Fibrillations
* Cardiac pathology or uncontrolled hypertension
* History of severe trauma/recent cervical surgery
* Uncontrolled systemic and inflammatory pathologies
* Congenital collagen compromise
* Presence of difficulties in performing the Initial Evaluation tests
* Language barriers
* Pending litigation or legal claim

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Only women older than 65 years with a pre-sarcopenia state are included.
Enrollment: 120 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Grip strength test | thirty weeks
  Accurate measurement of hand grip strength requires the use of a hand dynamometer (Jamar Plus) calibrated under well-defined (standardized) test conditions. Force values less than 16 Kg are considered positive.
Chair stand test | thirty weeks
  It can be used as an indicator of the strength of the lower limb muscles. It measures the amount of time a patient needs to get up five times from a sitting position without using their arms. It will help us to affirm that the person has a probable sarcopenia. Times greater than 15 seconds are considered positive

SECONDARY OUTCOMES:
SARC-F questionnaire | thirty weeks
  A simple questionnaire to rapidly diagnose sarcopenia with 5 questions for the initial detection of risk of sarcopenia (5 components: Strength, assistance in walking, rise from a chair, climb stairs, and falls). A score equal to or greater than 4 points better predicts the need for a more comprehensive evaluation.
Evaluation of changes in contraction velocity (m/s) | thirty weeks
  Velocity (m/s) of concentric contraction execution of a full extension of the lower limb will be evaluated to assess the changes in the force-velocity profile after performing the different interventions. It will be measured using the ADR linear encoder device and the mean value of five repetitions will be obtained.
Body Mass Index (BMI) | thirty weeks
  It is a measure used to assess a person's body weight in relation to their height. It is calculated by dividing a person's weight in kilograms by their height in meters squared (BMI = kg/m²).
Short Physical Performance Battery (SPPB) | thirty weeks
  Test to assess physical performance and degree of frailty consisting of 3 subtests: gait speed, balance, and lower limb strength. The maximum score is 12 points and a score ≤ 8 points indicates poor physical performance.
Gait speed | thirty weeks
  It is considered a fast, safe and very reliable test for sarcopenia, in a distance of 4 meters, values greater than 0.8 m/s are considered positive.
Timed Up and Go (TUG) | thirty weeks
  A predictive test for frailty and falls, where individuals are asked to get up from a standard chair, walk to a marker 3 m away, turn around, and sit down again. Times greater than 20 seconds are considered positive.
food frequency questionnaire (FFQ) | thirty weeks
  The 143-item questionnaire of the PREDIMED study, validated in Spain, was used to assess dietary habits. Nutrient intake was calculated using food composition tables, including values for macronutrients (protein, CHO, fat) and essential micronutrients (minerals and vitamins), each with the corresponding unit of measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salamanca, Salamanca, Spain

REFERENCES:
- [Derived] Polo-Ferrero L, Recio-Rodriguez JI, Gonzalez-Manzano S, Martin-Vallejo J, Barbero-Iglesias FJ, Montero-Errasquin B, Cruz-Jentoft AJ, Mendez-Sanchez R. Nutritional intake as a determinant of high-speed resistance and multicomponent training efficacy on strength in older women at risk of sarcopenia. A randomized clinical trial. Clin Nutr. 2025 Apr;47:103-111. doi: 10.1016/j.clnu.2025.02.015. Epub 2025 Feb 19. PMID 39999641
- [Derived] Polo-Ferrero L, Saez-Gutierrez S, Davila-Marcos A, Barbero-Iglesias FJ, Sanchez-Sanchez MC, Puente-Gonzalez AS, Mendez-Sanchez R. Effect of power training on function and body composition in older women with probable sarcopenia. A study protocol for a randomized controlled trial. PLoS One. 2025 Jan 6;20(1):e0313072. doi: 10.1371/journal.pone.0313072. eCollection 2025. PMID 39761305